CLINICAL TRIAL: NCT03510585
Title: Mucociliary Clearance, Airway Inflammation and Nasal Symptoms in Urban Motorcycle-drivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Naomi Kondo Nakagawa, Associate Professor of Faculdade de Medicina da Universidade de São Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP-FMUSP 221/11
Record Dates: First submitted 2013-06-18; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Attitude to Health
Keywords: mucociliary clearance; air pollution; nasal lavage; exhaled breath condensate; inflammation
MeSH Terms: conditions — Inflammation | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline and sniffing (Experimental): This RRC is the combination of positioning (laying down), sniffing (only one side), throat vibration and saline instillation. And then the other side.
  Interventions: Other: saline and sniffing
- sniffing (Placebo Comparator): Pacient will be in a lay down condition and will perform sniffing with throat vibration several times each side (but with no saline instillation)
  Interventions: Other: sniffing

INTERVENTIONS:
Other: saline and sniffing — This technique is a combination of positioning (laying down), saline instilation (5 ml in each side), sniffing (the side that received saline instilation) and throat vibration. Then the other side.
  Arms: saline and sniffing
Other: sniffing — This technique is a combination of positioning (laying down), sniffing (the side that received saline instilation) and throat vibration. Then the other side.
  Arms: sniffing

SUMMARY:
Professionals working in polluted areas may present increased airways symptoms and dysfunction. Rhinopharyngeal retrograde clearance (RRC) has been used to improve mucus clearance in infants with bronchitis and bronchiolitis. Flushing the nasal cavity with saline (S) has been used to reduce nasal inflammation in rhinitis and sinupathies. The aim of this study was to assess the effects of RRC and RRC plus S (RRC+S) on the airways in professional motorcyclists. Twenty-four male motorcyclists (mean age 36 years) were randomly assigned to RRC or RRC+S. Subjects were assessed at baseline and 15 days after interventions for airways assessments by saccharin test, mucus contact angle, cellularity in nasal lavage and airways symptoms with the use of SNOT-20 questionnaire. Data were analyzed by nonparametric ANOVA for repeated measures with Bonferroni´s correction. A passive nitrogen dioxide monitoring system was used to assess the mean personal air pollution exposure along the study period (NO2). The association between NO2 and the airways outcomes was analyzed by Spearman correlation test. At baseline, the two groups were similar in clinical, demographics and working aspects. From them, 100% had airways symptoms complaints and 33% had nasal MCC impairment. After treatments, both groups presented improvements in airways symptoms and nasal MCC. However, increased number of macrophages and ciliated cells were observed in nasal lavage of both groups. No associations between nitrogen dioxide and the outcome variables were detected. Rhinopharyngeal retrograde clearance seems to be useful in the clinical management of the upper airways symptoms and dysfunction in adults.

DETAILED DESCRIPTION:
The nonsmokers subjects aged 18 years to 45 years were enrolled in this study after agreement with the written informed consent. Subjects were randomly assigned to 15-days of one of the following interventions: RRC and RRC+S. Non pharmacological respiratory approaches may be useful in the management of the respiratory symptoms and dysfunctions air pollution-related. The purpose of this study was to determine whether saline instillation and/or retrograde rhinopharyngeal retrograde clearance are effective in the treatment of upper airways dysfunction through nasal mucociliary clearance, mucus properties, pH, cellularity and cytokines in nasal lavage and pH in exhaled breath condensate, as well as the airways symptoms (cough, wheeze, runny nose, hoarseness, among others) in motorcyclists due to urban air pollution.

ELIGIBILITY:
Inclusion Criteria:

* Professional motorcyclists aged 18 years to 45 years
* Agreement with the written informed consent

Exclusion Criteria:

* inability to understand and to follow commands,
* previous nasal surgery,
* respiratory infection in the previous 30 days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Nasal mucociliary clearance | 15 days
  Saccharine transit time test.

SECONDARY OUTCOMES:
Mucus physical properties | 15 days
  Contact angle

OTHER OUTCOMES:
Upper airway symptoms | 15 days
  Sinonasal Outcome Questionnaire -20

CONTACTS AND LOCATIONS:
Overall Officials: Paulo HN Saldiva, PhD, Study Director — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Faculdade de Medicina da Universidade de São Paulo, São Paulo

REFERENCES:
- [Result] Brant TC, Yoshida CT, Carvalho Tde S, Nicola ML, Martins JA, Braga LM, Oliveira RC, Leyton V, Andre CS, Saldiva PH, Rubin BK, Nakagawa NK. Mucociliary clearance, airway inflammation and nasal symptoms in urban motorcyclists. Clinics (Sao Paulo). 2014;69(12):867-70. doi: 10.6061/clinics/2014(12)13. PMID 25628001